CLINICAL TRIAL: NCT01456455
Title: Registry of Gastric Cancer and Brain Metastases
Brief Title: Gastric Cancer Metastasized to the Central Nervous System (CNS)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: UGICNS
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Gastric Cancer
Keywords: Central nervous system; pathological markers
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Descriptive registry to investigate frequency of HER-2 positive gastric cancer involving CNS.

Exploration of additional prognostic factors for brain involvement from gastric cancer.

DETAILED DESCRIPTION:
HER2 Status E-Cadherin Status

ELIGIBILITY:
Inclusion criteria:

* in order to be eligible for the study, the diagnosis of gastric cancer and/or lower esophageal cancer must be confirmed histologically. CNS involvement must be confirmed either via independent neuroradiological and/or positive CSF cytology.

Exclusion criteria:

* Patients whose diagnosis is not confirmed upon pathological review or where the CNS involvement cannot be confirmed after neuroradiological review will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: international
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-08; Primary Completion 2020-03 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
HER2 Status | 2 years
  Determination of HER2 Status on Tumor Tissue

SECONDARY OUTCOMES:
Outcome according to HER2 Status | 2 years

OTHER OUTCOMES:
Outcome according to ethnicity of patients | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Silvia Hofer, MD, Principal Investigator — University Hospital Zurich, Division of Oncology
Locations (1):
- Dept Oncology, University Hospital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feilchenfeldt J, Varga Z, Siano M, Grabsch HI, Held U, Schuknecht B, Trip A, Hamaguchi T, Gut P, Balague O, Khanfir K, Diebold J, Jochum W, Shoji H, Kushima R, Wagner D, Shimada Y, Cats A, Knuth A, Moch H, Aebi S, Hofer S. Brain metastases in gastro-oesophageal adenocarcinoma: insights into the role of the human epidermal growth factor receptor 2 (HER2). Br J Cancer. 2015 Sep 1;113(5):716-21. doi: 10.1038/bjc.2015.279. Epub 2015 Aug 27. PMID 26313663